CLINICAL TRIAL: NCT05836012
Title: A Phase 2, Multi-country, Randomized, Double-blind, Placebo-controlled Trial to Evaluate Safety and Immunogenicity When HIL-214 is Concomitantly Administered With Routine Pediatric Vaccines in Healthy Infants
Brief Title: Safety and Immunogenicity of HIL-214 With Routine Pediatric Vaccines
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: HilleVax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-206
Record Dates: First submitted 2023-03-21; First posted 2023-05-01 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): HIL-214 (1 dose at 4 months of age and 1 dose at 6 months of age) and routine childhood vaccines according to schedule.
  Interventions: Biological: HIL-214
- Placebo (Placebo Comparator): Placebo (1 dose at 4 months of age and 1 dose at 6 months of age) and routine childhood vaccines according to schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HIL-214 — 2 injections - given at 4 months and the second at 6 months of age.
  Arms: Experimental
Biological: Placebo — 2 injections - given at 4 months and the second at 6 months of age.
  Arms: Placebo

SUMMARY:
This is a phase 2, multi-country, randomized, double-blind, placebo-controlled trial to evaluate the immune response to routine pediatric vaccinations when co-administered with HIL-214 or placebo in healthy infants. This trial will also evaluate the safety profile of a 2-dose regimen of HIL-214 co-administered with routine pediatric vaccines.

DETAILED DESCRIPTION:
Epidemiologic studies have shown that gastroenteritis in infants is associated with several viruses, including norovirus, sapovirus and rotavirus. These viruses together or individually can be associated with illness ranging from asymptomatic to serious. Asymptomatic infection can create a reservoir, allowing further spread of the virus, whereas serious illness can lead to death, particularly in the very young, very old or immunocompromised. As the burden of rotavirus in children decreases due to successful rotavirus vaccination programs in infants, norovirus infections are increasingly recognized as the primary cause of acute gastroenteritis (AGE) in many countries around the world. Currently, there is no available vaccine to counter the disease burden associated with norovirus. Vaccinating at an early age would reduce the severe illness in young children and also reduce the asymptomatic cases which act as a vehicle for transmission within the population. As infants already receive multiple vaccines during the first months of life, an additional vaccination must fit into the immunization scheme in a convenient way for compliance. It must also have an acceptable safety profile and be immunogenic without interfering with the immune response to routine childhood vaccines.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged 2 months (+14 days).
* Male or female.
* Infants who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
* The subject's LAR signs and dates a written, informed consent form (ICF) and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
* Infants whose LARs can and are willing to comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

* Clinically significant abnormality in growth by height, weight, or head circumference (according to local guidelines).
* Gastrointestinal abnormalities or any chronic gastrointestinal disease, including any uncorrected congenital malformation of the gastrointestinal tract according to medical history and/or physical examination.
* Known hypersensitivity or allergy to any of the investigational vaccine components (including excipients).
* Severe reaction to routine childhood vaccine(s) administered at Visit 1.
* Any clinically significant active infection (as assessed by the investigator) or temperature

  ≥38.0°C (>100.4°F), within 3 days of intended trial vaccination.
* Any serious chronic or progressive disease according to the judgment of the investigator (e.g., cardiac, renal or hepatic disease).
* Individuals with history of, e.g., convulsions/febrile convulsions, or any illness, that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the subjects due to participation in the trial.
* Known or suspected impairment/alteration of immune function.
* Subjects with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Subjects who received or are scheduled to receive any licensed or authorized vaccines not planned in this trial within 14 days (for inactivated vaccines) or within 28 days (for live vaccines) before or after any dose of trial vaccine. Note: Flu and/or COVID vaccine can be administered per local guidelines at any time during the trial.
* Subjects participating in any clinical trial with another investigational product 30 days prior to first trial visit or due to participate in another clinical trial at any time during the conduct of this trial.
* Subjects known to be positive for or in evaluation for possible human immunodeficiency virus infection.
* Subject's LAR or subject's first-degree relatives involved in the trial conduct.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 329 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - Velocity Clinical Research - Lafayette, Lafayette, Louisiana
  - Boeson Research MSO, Missoula, Montana
  - Velocity Clinical Research - Hastings, Hastings, Nebraska
  - Frontier Pediatric Care, Lincoln, Nebraska
  - La Providence Pediatrics Clinic - Chemidox Clinical Trials (Hypercore), Houston, Texas
  - Alliance for Multispecialty Research LLC - Kaysville, Kaysville, Utah
  - Alliance for Multispecialty Research LLC - Syracuse, Syracuse, Utah
- Panama (3):
  - CEVAXIN-La Chorrera, La Chorrera
  - Cervaxin-Avenida Mexico, Panama City
  - Cervaxin-Tocumen, Panama City
- Puerto Rico (2):
  - BRCR Global, San Juan
  - HACTR, San Juan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the trial at 10 investigative sites in Panama and the United States from 10 June 2023 to 08 July 2024.
Pre-assignment Details: Participants were enrolled in 1 of 2 treatment arms and received 2 doses of either HIL-214, a norovirus vaccine comprising 50 µg GI.1 virus-like particle (VLP) and 150 µg GII.4c VLP, adjuvanted with 500 µg of aluminum hydroxide, or placebo.
Groups:
- Placebo: 1 dose of placebo at 4 months of age and 1 dose of placebo at 6 months of age, and routine childhood vaccines according to schedule.
- HIL-214: 1 dose of HIL-214 at 4 months of age and 1 dose of HIL-214 at 6 months of age, and routine childhood vaccines according to schedule.
Period: Overall Study
Arm/Group | Placebo | HIL-214
Started | 164 | 165
Completed | 160 | 161
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Reason not included in pre-specified categories | 2 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set; All participants that were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | HIL-214 | Total
Number analyzed (Participants) | 164 | 165 | 329
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 164 | 165 | 329
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 125.7 (4.35) | 125.6 (4.48) | 125.7 (4.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 82 | 164
  Male | 82 | 83 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 159 | 160 | 319
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaskan Native | 1 | 0 | 1
  Race/Ethnicity: Black or African American | 2 | 1 | 3
  Race/Ethnicity: White | 9 | 9 | 18
  Race/Ethnicity: More than one race | 151 | 154 | 305
  Race/Ethnicity: Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
  Panama | 150 | 152 | 302
Prior Vaccinations [Count of Participants; unit: Participants]
  Yes | 163 | 161 | 324
  No | 1 | 4 | 5
Breastfeeding Status [Count of Participants; unit: Participants]
  Breastfeeding | 143 | 146 | 289
  Not breastfeeding | 21 | 19 | 40
Weight [Mean (Standard Deviation); unit: kg] | 7.00 (0.892) | 7.01 (0.877) | 7.00 (0.883)
Length [Mean (Standard Deviation); unit: cm] | 61.84 (2.221) | 62.12 (2.219) | 61.98 (2.221)
Head Circumference [Mean (Standard Deviation); unit: cm] | 41.24 (1.217) | 41.33 (1.290) | 41.29 (1.253)

OUTCOME MEASURES:

1. Primary Outcome: Immune Response to the Licensed Pediatric DTaP-Hib-IPV-HepB Vaccine Co-administered With a 2-dose Regimen of HIL-214 at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo.
Description: Evaluate the immune response to the licensed pediatric DTaP-Hib-IPV-HepB vaccine co-administered with a 2-dose regimen of HIL-214 at 4 and 6 months of age, compared to that of the routine pediatric vaccine co-administered with placebo. Due to differing local availability of licensed DTaP-Hib-IPV-HepB vaccine, data are presented by country (Panama and USA).
  Outcome measures:
  * Binary (yes/no) variable indicating anti-DT immunoglobulin G (IgG) concentration ≥0.1 IU/mL.
  * Binary variable indicating anti-TT IgG concentration ≥0.1 IU/mL.
  * Anti-pertussis [FHA], [PRN] and [PTX]) IgG concentrations.
  * Binary variable indicating anti-poliovirus neutralizing antibody titers ≥1:8,
  * Binary variable indicating anti-Haemophilus influenzae type b
  * Binary variable indicating anti-hepatitis b surface antigen
  Geometric mean (geometric mean standard deviation) anti-FHA, anti-PRN, and anti-PTX are presented as a separate outcome.
Time Frame: 28 days post-dose 2
Population: Immunology Evaluable Analysis Set; all participants in the randomized analysis set that received all doses of all study vaccines (routine and trial vaccines) within the required time window.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (Panama); Placebo (USA): 1 dose of placebo at 4 months of age and 1 dose of placebo at 6 months of age, and routine childhood vaccines according to schedule.
- HIL-214 (Panama); HIL-214 (USA): 1 dose of HIL-214 at 4 months of age and 1 dose of HIL-214 at 6 months of age, and routine childhood vaccines according to schedule.
Arm/Group | Placebo (Panama) | HIL-214 (Panama) | Placebo (USA) | HIL-214 (USA)
Number analyzed (Participants) | 147 | 139 | 9 | 9
percentage of participants
  Anti-diphtheria toxoid IgG concentration ≥0.1 IU/mL. | 99.3 | 100 | 100 | 100
  Anti-tetanus toxoid IgG concentration ≥0.1 IU/mL | 100 | 100 | 100 | 100
  Anti-poliovirus type 1 neutralizing antibody titers ≥3 log2: number analyzed (Participants) | 145 | 130 | 6 | 6
  Anti-poliovirus type 1 neutralizing antibody titers ≥3 log2 | 100 | 100 | 100 | 83.3
  Anti-poliovirus type 2 neutralizing antibody titers ≥3 log2: number analyzed (Participants) | 145 | 130 | 6 | 6
  Anti-poliovirus type 2 neutralizing antibody titers ≥3 log2 | 100 | 100 | 100 | 100
  Anti-poliovirus type 3 neutralizing antibody titers ≥3 log2: number analyzed (Participants) | 145 | 130 | 6 | 6
  Anti-poliovirus type 3 neutralizing antibody titers ≥3 log2 | 99.3 | 99.2 | 100 | 100
  Anti-PRP IgG concentration ≥ 0.15 ug/mL | 100 | 100 | 100 | 100
  Anti-HBsAg IgG concentration ≥10 mIU/mL: number analyzed (Participants) | 147 | 139 | 8 | 8
  Anti-HBsAg IgG concentration ≥10 mIU/mL | 100 | 100 | 100 | 100

2. Primary Outcome: Immune Response to the Licensed Pediatric DTaP-Hib-IPV-HepB Vaccine Co-administered With a 2-dose Regimen of HIL-214 at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo.
Description: Evaluate the immune response to the licensed pediatric DTaP-Hib-IPV-HepB vaccine co-administered with a 2-dose regimen of HIL-214 at 4 and 6 months of age, compared to that of the routine pediatric vaccine co-administered with placebo. Due to differing local availability of licensed DTaP-Hib-IPV-HepB vaccine, data are presented by country (Panama and USA).
  Outcome measures:
  Geometric mean anti-FHA, anti-PRN, and anti-PTX concentrations
Time Frame: 28 days post-dose 2
Population: Immunology Evaluable Analysis Set; all participants in the randomized analysis set that receive all doses of all study vaccines (routine and trial vaccines) within the required time window.
Measure: Geometric Mean (Standard Deviation); unit: IU/mL
Arm/Group | Placebo (Panama) | HIL-214 (Panama) | Placebo (USA) | HIL-214 (USA)
Number analyzed (Participants) | 147 | 139 | 9 | 9
IU/mL
  Anti-pertussis FHA concentration | 83.958 (1.8338) | 78.726 (1.8566) | 32.515 (2.9346) | 26.358 (2.7499)
  Anti-pertactin (PRN) concentration | 92.605 (2.1811) | 84.617 (2.2496) | 61.222 (2.6526) | 43.417 (2.7743)
  Anti-pertussis toxin (PTX) concentration | 48.536 (1.8552) | 48.906 (2.0150) | 80.713 (2.2249) | 43.066 (2.5144)

3. Primary Outcome: Immune Response to the Licensed Pediatric Pneumococcal 13 Valent (PCV13) Vaccine Co-administered With a 2-dose Regimen of HIL-214 at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo.
Description: The outcome was assessed using measurements of immune response to the concomitant anti-pneumococcal capsular polysaccharide IgG [serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F, 18C, and 23F]) at 28 days post-dose. Geometric mean concentrations are presented.
Time Frame: 28 days post-dose 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 154 | 143
ug/mL
  Anti-pneumococcal IgG concentration for serotype 1 | 5.255 (1.9827) | 5.802 (2.2008)
  Anti-pneumococcal IgG concentration for serotype 3 | 0.777 (2.3728) | 0.747 (2.2117)
  Anti-pneumococcal IgG concentration for serotype 4 | 2.958 (1.8468) | 2.773 (2.0253)
  Anti-pneumococcal IgG concentration for serotype 5 | 2.378 (1.9223) | 2.429 (1.9277)
  Anti-pneumococcal IgG concentration for serotype 6A | 7.660 (2.0384) | 7.414 (2.2194)
  Anti-pneumococcal IgG concentration for serotype 6B | 6.419 (2.3854) | 5.459 (2.7604)
  Anti-pneumococcal IgG concentration for serotype 7F | 5.091 (1.6726) | 5.063 (1.7727)
  Anti-pneumococcal IgG concentration for serotype 9V | 3.881 (1.9259) | 3.568 (2.1651)
  Anti-pneumococcal IgG concentration for serotype 14: number analyzed (Participants) | 154 | 142
  Anti-pneumococcal IgG concentration for serotype 14 | 11.819 (2.3158) | 12.017 (2.3278)
  Anti-pneumococcal IgG concentration for serotype 19A | 3.203 (2.0635) | 3.069 (1.9742)
  Anti-pneumococcal IgG concentration for serotype 19F | 5.822 (2.0030) | 5.487 (2.1713)
  Anti-pneumococcal IgG concentration for serotype 18C | 2.997 (1.8435) | 3.040 (1.9344)
  Anti-pneumococcal IgG concentration for serotype 23F | 2.885 (2.5878) | 2.543 (2.7745)

4. Primary Outcome: Immune Response to the Licensed Pediatric Rotavirus Vaccine (RV1) Vaccine Co-administered With a 2-dose Regimen of HIL-214 at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo.
Description: This outcome was assessed using measurements of immune response to the concomitant RV1 vaccine (anti-RV1 IgA). Geometric mean concentrations at 28 days post-dose 2 are reported.
Time Frame: 28 days post-dose 2
Population: Immunology Evaluable Analysis Set, all participants in the randomized analysis set that receive all doses of all study vaccines (routine and trial vaccines) within the required time window
Measure: Geometric Mean (Standard Deviation); unit: U/mL
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 155 | 147
U/mL | 67.772 (4.0633) | 87.694 (4.2618)

5. Secondary Outcome: Immunogenicity of a 2-dose Regimen of HIL-214 Co-administered With Routine Pediatric Vaccines at 4 and 6 Months of Age.
Description: Anti-norovirus (GI.1 and GII.4c) HBGA-blocking antibodies were measured at prior to dose 1 (~4 months of age) and 28 days post-dose 2 (~6 months of age). Seroresponse was defined as a fold increase from baseline greater than or equal to 4. Seroresponse rates and 95% confidence intervals (CIs) are presented. Data are stratified by country (Panama and USA).
Time Frame: Pre-dose 1 and 28 days post-dose 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo (USA): 1 dose of placebo at 4 months of age and 1 dose of placebo at 6 months of age and routine childhood vaccines according to schedule
- HIL-214 (USA): 1 dose of HIL-214 at 4 months of age and 1 dose of HIL 214 at 6 months of age and routine childhood vaccines according to schedule.
Arm/Group | Placebo (Panama) | HIL-214 (Panama) | Placebo (USA) | HIL-214 (USA)
Number analyzed (Participants) | 123 | 119 | 6 | 7
percentage of participants
  Anti-GI.1 seroresponse by HBGA-blocking assay at 28 days post-dose 2: number analyzed (Participants) | 123 | 118 | 6 | 7
  Anti-GI.1 seroresponse by HBGA-blocking assay at 28 days post-dose 2 | 4.1 [1.3 to 9.2] | 97.5 [92.7 to 99.5] | 0 [0.0 to 45.9] | 100 [59.0 to 100]
  Anti-GII.4c seroresponse by HBGA-blocking assay at 28 days post-dose 2: number analyzed (Participants) | 122 | 119 | 6 | 7
  Anti-GII.4c seroresponse by HBGA-blocking assay at 28 days post-dose 2 | 1.6 [0.2 to 5.8] | 51.3 [41.9 to 60.5] | 0 [0.0 to 52.5] | 16.7 [0.4 to 64.1]
  Anti-GI.1 and GII.4c seroresponse by HBGA-blocking assay at 28 days post-dose 2: number analyzed (Participants) | 121 | 115 | 5 | 6
  Anti-GI.1 and GII.4c seroresponse by HBGA-blocking assay at 28 days post-dose 2 | 0.8 [0.0 to 4.5] | 53.0 [43.5 to 62.4] | 0 [0.0 to 52.2] | 16.7 [0.4 to 64.1]

6. Secondary Outcome: Evaluate the Safety Profile of a 2-dose Regimen of HIL-214 Co-administered With Routine Pediatric Vaccines at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo.
Description: Percentage of participants with solicited local (injection site) reactions within 7 days of any vaccine administration. Assessed reactions included pain, redness, induration, and swelling.
Time Frame: Day 1 to Day 7 post-dose 1 and Day 1 to Day 7 post-dose 2
Population: Safety Analysis Set, all participants that received trial vaccine (HIL-214 or placebo)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 164 | 165
percentage of participants | 38.4 | 41.2

7. Secondary Outcome: Evaluate the Safety Profile of a 2-dose Regimen of HIL-214 Co-administered With Routine Pediatric Vaccines at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo.
Description: Percentage of participants with solicited systemic adverse events (AEs) within 7 days of any vaccine administration. Assessed AEs included drowsiness, irritability/fussiness, loss of appetite, fever, vomiting, and diarrhea.
Time Frame: Day 1 to Day 7 post-dose 1 and Day 1 to Day 7 post-dose 2
Population: Safety Analysis Set; all participants that received trial vaccine (HIL 214 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 164 | 165
percentage of participants | 54.9 | 46.1

8. Secondary Outcome: Evaluate the Safety Profile of a 2-dose Regimen of HIL-214 Co-administered With Routine Pediatric Vaccines at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo.
Description: Percentage of participants with adverse events (AEs) leading to vaccine discontinuation or trial withdrawal.
Time Frame: Day 1 to 28 days post-dose 1 (vaccine discontinuation); Day 1 to 12 months post-dose 1
Population: Safety Analysis Set; all participants that received trial vaccine (HIL-214 or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 164 | 165
percentage of participants
  AE leading to vaccine discontinuation | 0 | 0
  AE leading to trial withdrawal | 0 | 0

9. Secondary Outcome: Evaluate the Safety Profile of a 2-dose Regimen of HIL-214 Co-administered With Routine Pediatric Vaccines at 4 and 6 Months of Age, Compared to That of the Routine Pediatric Vaccines Co-administered With Placebo
Description: Percentage of participants with medically attended adverse events (AEs) at any point during the trial.
Time Frame: Day 1 to 12 months post-dose 1
Population: Safety Analysis Set; all participants that received trial vaccine (HIL-214 or placebo)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 164 | 165
percentage of participants | 63.4 | 65.5

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from Day 1 to 12 months post-dose 1; unsolicited adverse events were assessed for up to 28 days post-dose 1 and 28 days post-dose 2.
Groups:
- Placebo: 1 dose of placebo at 4 months of age and 1 dose of placebo at 6 months of age), and routine childhood vaccines according to schedule.
- HIL-214: 1 dose of HIL-214 at 4 months of age and 1 dose of HIL-214 at 6 months of age), and routine childhood vaccines according to schedule.
Arm/Group | Placebo | HIL-214
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/165
Serious Adverse Events (participants affected / at risk) | 7/164 | 3/165
Other Adverse Events (participants affected / at risk) | 81/164 | 77/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=164) | HIL-214 (N=165)
Bronchiolitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia respiratory syncytial virus (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=164) | HIL-214 (N=165)
Nasopharyngitis (Infections and infestations) | 64 | 55
Gastroenteritis (Infections and infestations) | 5 | 10
Bronchiolitis (Infections and infestations) | 4 | 8
Pyrexia (General disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT05836012/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT05836012/SAP_001.pdf